CLINICAL TRIAL: NCT02564640
Title: Comparison of Hemodynamic Changes After Endotracheal Intubation by Using the Videolaryngoscope and the Macintosh Direct Laryngoscope in Elderly Hypertensive Patients
Brief Title: Comparison of Hemodynamic Changes by Using the Videolaryngoscope and the Macintosh Laryngoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AntalyaTRH 008
Record Dates: First submitted 2015-09-28; First posted 2015-10-01 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-06

CONDITIONS: Anesthesia Intubation Complication
Keywords: videolaryngoscope; direct laryngoscope; hemodynamic changes; elderly patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- videolaryngoscope (Active Comparator): patients intubated by using the videolaryngoscopy
  Interventions: Device: videolaryngoscope
- Macintosh laryngoscope (Active Comparator): patients intubated by using the Macintosh laryngoscope
  Interventions: Device: Macintosh laryngoscope

INTERVENTIONS:
Device: videolaryngoscope — patients intubated by using the videolaryngoscope
  Arms: videolaryngoscope
Device: Macintosh laryngoscope — patients intubated by using the Macintosh laryngoscope
  Arms: Macintosh laryngoscope

SUMMARY:
Tracheal intubation techniques that avoid or minimize pharyngolaryngeal stimulation might attenuate the hemodynamic stress response. Tracheal intubation using video laryngoscope needs comparatively less airway manipulation so, the investigators expect less hemodynamic response while using videolaryngoscope.

DETAILED DESCRIPTION:
The hemodynamic stress response to tracheal intubation can precipitate adverse cardiovascular events in patients with cardiovascular disease. Which is shown to greatly increase the risk of myocardial infarction or stroke, especially in elderly patients with hypertension. Direct laryngoscopy and laryngoscopic stimulation of pharyngolaryngeal structures may be an important factor in the hemodynamic stress response associated with tracheal intubation.

Patients were randomly allocated to two groups using a permuted block randomization method: 1) patients intubated by using the videolaryngoscopy 2) patients intubated by using the Macintosh laryngoscope . SAP, MAP, and heart rate were measured and recorded in the operating room: At baseline, before intubation, immediately after intubation and 1,2,3,4 and 5 minutes after tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status II-III,
* aged over 65 years,
* controlled hypertensive patients,
* scheduled for elective coronary artery bypass grafting.

Exclusion Criteria:

* American Society of Anesthesiologists Physical Status IV,
* ejection fraction < 40%,
* any anatomical abnormality in head, neck or face,
* Mallampati score of IV,
* history of difficult intubation or laryngoscopy

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Blood pressure changes during tracheal intubation ( mmHg ) , | At baseline, 1 minute before intubation, and 1,2,3,4 and 5 minutes after tracheal intubation

SECONDARY OUTCOMES:
Heart rate changes during tracheal intubation (beats per minute) | At baseline, 1 minute before intubation, and 1,2,3,4 and 5 minutes after tracheal intubation
ST segment elevation in electrocardiogram indicating myocardial ischaemia during tracheal intubation | At baseline, 1 and 5 minutes after tracheal intubation.
  During tracheal intubation electrocardiogram is monitorized.
Arrhythmic changes in electrocardiogram during tracheal intubation | At baseline, 1 and 5 minutes after tracheal intubation.
  During tracheal intubation electrocardiogram is monitorized.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgun Kavrut Ozturk, MD, Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Kihara S, Brimacombe J, Yaguchi Y, Watanabe S, Taguchi N, Komatsuzaki T. Hemodynamic responses among three tracheal intubation devices in normotensive and hypertensive patients. Anesth Analg. 2003 Mar;96(3):890-895. doi: 10.1213/01.ANE.0000048706.15720.C9. PMID 12598280
- [Background] Kanaide M, Fukusaki M, Tamura S, Takada M, Miyako M, Sumikawa K. Hemodynamic and catecholamine responses during tracheal intubation using a lightwand device (Trachlight) in elderly patients with hypertension. J Anesth. 2003;17(3):161-5. doi: 10.1007/s00540-003-0166-8. PMID 12911202
- [Result] Xue FS, Zhang GH, Li XY, Sun HT, Li P, Li CW, Liu KP. Comparison of hemodynamic responses to orotracheal intubation with the GlideScope videolaryngoscope and the Macintosh direct laryngoscope. J Clin Anesth. 2007 Jun;19(4):245-50. doi: 10.1016/j.jclinane.2006.11.004. PMID 17572317
- [Result] Xue FS, Zhang GH, Li XY, Sun HT, Li P, Sun HY, Xu YC, Liu Y. Comparison of haemodynamic responses to orotracheal intubation with GlideScope videolaryngoscope and fibreoptic bronchoscope. Eur J Anaesthesiol. 2006 Jun;23(6):522-6. doi: 10.1017/S0265021506000299. Epub 2006 Mar 1. PMID 16507195